CLINICAL TRIAL: NCT07289815
Title: Construction and Application of an Intelligent Collaborative Cardiac Rehabilitation Management Model for Young and Middle-aged Patients With Myocardial Infarction Based on Intervention Mapping
Brief Title: Construction and Application of an Intelligent Collaborative Cardiac Rehabilitation App for Middle-aged and Young Patients With Myocardial Infarction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-302
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction; Cardiac Rehabilitation; APP
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group, On the basis of conventional rehabilitation guidance, the "Cardiac Rehabilitatio (Experimental)
  Interventions: Behavioral: Cardiac Rehabilitation Management App
- normal group, conventional rehabilitation guidance (Active Comparator)
  Interventions: Behavioral: Conventional Rehabilitation Guidance

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation Management App — Develop a targeted and actionable health management APP focusing on five major health issues (diet, medication, exercise, psychology, and smoking cessation). The experimental group will use it for check-in, while the APP will be equipped with a management mechanism, and the intervention will last for 6 months.
  Arms: experimental group, On the basis of conventional rehabilitation guidance, the "Cardiac Rehabilitatio
Behavioral: Conventional Rehabilitation Guidance — ① Before discharge, cardiologists will provide face-to-face health education to patients, covering the rehabilitation goals of myocardial infarction (MI), risk factor control, dietary recommendations, exercise precautions, medication adherence, and prevention of common complications.② Patients will be given a uniformly compiled printed Cardiac Rehabilitation Guidance Manual for self-directed reading and learning.③ After discharge, the responsible nurse will conduct health follow-ups via phone call or WeChat at the 1st week, 1st month, 3rd month, and 6th month to monitor rehabilitation progress and medication compliance, and provide targeted guidance.
  Arms: normal group, conventional rehabilitation guidance

SUMMARY:
This study is guided by the intervention mapping theory, combined with Fogg's behavior model and digital health technologies, focusing on the key rehabilitation obstacles and behavioral characteristics of young and middle-aged MI patients. It constructs a "smart + collaborative" out-of-hospital rehabilitation management model. This model, through systematic needs assessment and problem logical modeling [11], develops individualized rehabilitation paths covering multiple dimensions of intervention such as exercise, diet, medication, and psychological regulation. It relies on digital means such as mobile terminals, online education, behavior check-ins, real-time feedback, and remote follow-ups to achieve intelligent rehabilitation management. At the same time, it emphasizes the multi-disciplinary collaboration mechanism, integrating team members from cardiology, nursing, nutrition, rehabilitation, and psychology, forming a collaborative work system with information sharing, task complementarity, and consistent goals. Together, they promote the activation of patient motivation, improvement of behavioral ability, and improvement of rehabilitation compliance. The study will also verify its feasibility and initial effects in a real clinical environment, and evaluate its practical value in improving rehabilitation behaviors, promoting functional recovery, and enhancing quality of life. This study not only innovatively integrates intervention mapping and behavioral science models into the rehabilitation management of young and middle-aged MI patients in theory, filling the gap in existing rehabilitation models for this group, but also explores the path of digital rehabilitation intervention that can be promoted and replicated in grassroots clinical practice. The research results can provide practical basis for the construction of the smart rehabilitation service system under the background of "Healthy China 2030", and have important practical significance and social value.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Ward 1 were assigned to the intervention group, and patients in Ward 2 served as the control group. The inclusion criteria were as follows: ① aged 18-60 years; ② diagnosed by cardiologists as meeting the clinical diagnostic criteria for myocardial infarction (MI) established by the Cardiology Branch of the Chinese Medical Association; ③ having basic smartphone operation skills to use the App normally; ④ providing informed consent and signing the research consent form.

Exclusion Criteria:

* ① Complicated with severe hepatic or renal insufficiency, malignant tumors, cognitive impairment, or mental illnesses; ② Patients with NYHA class Ⅳ or definite exercise contraindications (e.g., those assessed as high-risk in exercise risk evaluation) who are unable to participate in exercise prescription intervention; ③ Patients who have difficulty completing follow-up or withdraw midway.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Condition of Cardiac Function Recovery | Assessments will be conducted at four time points: before the intervention (T0), 1 month after the intervention (T1), 3 months after the intervention (T2), and 6 months after the intervention (T3).
  It is evaluated by the 6-minute walk distance (6MWD, six minutes walk test).

OTHER OUTCOMES:
Quality of Life (QoL) | Assessments will be conducted at four time points: before the intervention (T0), 1 month after the intervention (T1), 3 months after the intervention (T2), and 6 months after the intervention (T3).
  The Chinese version of the Seattle Angina Questionnaire (SAQ) [37] was used to assess patients' health-related quality of life over the past 4 weeks.
Patient Satisfaction | It will be distributed at three time points: 1 month after the intervention (T1), 3 months after the intervention (T2), and 6 months after the intervention (T3).
  A self-designed questionnaire on App usage satisfaction will be used, covering 6 dimensions: interface friendliness, function practicality, personalization level, interactive experience, overall satisfaction, and recommendation willingness.
Self-Management Ability Score | Assessments will be conducted at four time points: before the intervention (T0), 1 month after the intervention (T1), 3 months after the intervention (T2), and 6 months after the intervention (T3).
  The Chinese Self-Management Scale (CSMS) was used for assessment, which includes 3 dimensions (daily life management, disease medical management, and emotional cognitive management) with a total of 27 items.

IPD SHARING:
Plan to Share IPD: No